CLINICAL TRIAL: NCT00156871
Title: Individualized Exercise Program for Treatment of Fatigue in Patients After Hematologic Stem Cell Transplant
Brief Title: Individualized Exercise Program for Treatment of Fatigue in Patients After Hematologic Stem Cell Transplant (HSCT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alberta Health services (Other)
Collaborators: Alberta Cancer Foundation (Other)
Organization: AHS Cancer Control Alberta (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 181710-DRD 16; ACF 717905155
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2011-08

CONDITIONS: Fatigue
Keywords: transplant; fatigue; exercise; Malignant disease
MeSH Terms: conditions — Fatigue; Motor Activity | interventions — Exercise

INTERVENTIONS:
Behavioral: exercise

SUMMARY:
The purpose of this study is to investigate the impact of fatigue in severely affected transplant patients.

DETAILED DESCRIPTION:
Investigates impact of a monitored program in kinesiology lab at the University of Calgary on fatigue in severely affected transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Severe fatigue post transplant

Exclusion Criteria:

* Other conditions contributing to fatigue (graft versus host disease)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2003-04; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Fatigue score

CONTACTS AND LOCATIONS:
Overall Officials: James Russell, Study Director — AHS Cancer Control Alberta; Nicole Colos-Reed, Phd, Principal Investigator — University of Calgary
Locations (1):
- Tom Baker Cancer Centre, Calgary, Alberta, Canada